CLINICAL TRIAL: NCT00651014
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Ezetimibe 10 mg or Placebo Co-administered With Existing Simvastatin 10mg or 20mg in Attaining Low-Density Lipoprotein Cholesterol Target Levels in Patients With Hypercholesterolemia and Coronary Heart Disease and/or Type II Diabetes
Brief Title: Ezetimibe Plus Simvastatin Versus Simvastatin in Patients With Hypercholesterolemia and Coronary Risk Factors (P03405)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow subject recruitment and lack of medical and scientific merit due to change in new standard of therapy during that same period.
Sponsor: Organon and Co (Industry)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03405
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Atherosclerosis
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ezetimibe (Experimental)
  Interventions: Drug: Ezetimibe
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ezetimibe — oral tablet; ezetimibe 10 mg once daily for 6 weeks (added to ongoing simvastatin 10 or 20 mg once daily)
  Other Names: SCH 58235; Zetia
  Arms: Ezetimibe
Drug: Placebo — oral tablet; ezetimibe placebo once daily for 6 weeks (added to ongoing simvastatin 10 or 20 mg once daily)
  Arms: Placebo

SUMMARY:
The study was designed to assess whether 6 weeks of co-administration of ezetimibe and simvastatin is more effective than simvastatin monotherapy in allowing patients in the CHD risk strata of the NCEP III guidelines to achieve their LDL-C target goal of <=3.0 mmol/L. As this study was to be conducted in Canada, the target LDL-C goal for patients with CHD, or type II diabetic patients >30 years old with no CHD, was <2.5 mmol/L.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age and treated with simvastatin 10 mg or 20 mg for at least 6 weeks and LDL-C levels of > 2.5 mmol/L to <=4.20 mmol/L (97 mg/dL to 160 mg/dL) at Visit 1.
* history of coronary heart disease (type II diabetic patients > 30 years old with no CHD)
* triglycerides <= 4.00 mmol/L drawn, and liver transaminases (ALT, AST) <=50% above the upper limit of normal at Visit 2, with no active liver disease, and/or creatine kinase (CK) <=50% above the upper limit of normal

Exclusion Criteria:

* subjects with Body Mass Index >=35 kg/sqm at Visit 1
* alcohol consumption > 14 drinks per week
* pregnant or lactating
* treated with any other investigational drug within 30 days prior Visit 1
* previously treated with ezetimibe or participated in a clinical study with ezetimibe
* any condition or situation which, in the opinion of the investigator, might pose a risk to the patient or interfere with participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching LDL-C goal of < 2.5 mmol/L (97 mg/dL) at endpoint. | 6 weeks

SECONDARY OUTCOMES:
Percent change from baseline to endpoint in LDL-C. | 6 weeks
Percent change from baseline to endpoint in total cholesterol (TC) triglycerides, HDL-C, non-HDL-C, LDL-C/HDL-C ratio, TC/HDL-C ratio, and apolipoprotein B. | 6 weeks
Safety/tolerability: adverse events, laboratory test results, vital signs. | Throughout study